CLINICAL TRIAL: NCT04874558
Title: Novel Ultra-low-dose Chest CT Technique to Screen for Pulmonary Arteriovenous Malformations in Pediatric Patients With Hereditary Hemorrhagic Teleangiectasia
Brief Title: Ultra-low-dose Chest CT for HHT
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nadir Demirel, Principal Investigator, Mayo Clinic
Other Study IDs: 21-000324
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Low-dose contrast-enhanced chest CT exam: Subjects will undergo a low-dose contrast-enhanced chest CT exam with coverage from the neck base through the lungs to the upper abdomen on a third-generation dual-source CT scanner as part of their routine clinical visit based on current guidelines.
  Interventions: Diagnostic Test: Ultra-low dose chest CT

INTERVENTIONS:
Diagnostic Test: Ultra-low dose chest CT — A novel CT technique with a new dose optimization and efficiency technology and automatic kV selection, which greatly reduces the dose of radiation exposure compared to a standard chest CT.

SUMMARY:
This study aims to develop a novel ultra-low dose chest CT technology for use in Hereditary Hemorrhagic Teleangiectasia (HHT) patients and to determine the lowest possible radiation dose that is achievable without sacrificing the diagnostic quality.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1 to 17 years
* Diagnosed with positive HHT causing mutations or based on Curacao criteria

Exclusion Criteria:

* Acute respiratory distress
* Unstable cardiovascular status
* Pneumothorax, hemoptysis
* Pulmonary edema
* Pulmonary emboli
* Fractured ribs or other chest trauma
* Recent bronchoscopy
* Lung transplantation

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients followed by HHT clinic who are ordered a chest CTA.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultra-low dose images PAVM detection | Baseline
  Number of images detecting PAVM using the ultra-low dose images (50% or lower compared to the full dose)

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Demirel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No